CLINICAL TRIAL: NCT01977287
Title: A Pilot Study to Assess the Effects of Using FES or AFO as an Assistive Mobility for Period of 12 Weeks for People With Multiple Sclerosis With Foot Drop
Brief Title: Walking With FES or AFO in People With MS With Foot Drop
Status: Completed | Type: Observational
Sponsor: Queen Margaret University (Other)
Collaborators: Multiple Sclerosis Society UK (Unknown); NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Marietta van der Linden, Dr, Queen Margaret University
Other Study IDs: FESvsAFO2013
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis; Foot Drop
Keywords: Multiple Sclerosis; Functional Electrical Stimulation; Ankle Foot Orthosis; Walking performance; gait analysis; fatigue; activity monitoring
MeSH Terms: conditions — Multiple Sclerosis; Peroneal Neuropathies; Fatigue | interventions — Splints

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Functional Electrical Stimulation: The Functional Electrical Stimulation (FES) group will be asked to use their clinically prescribed FES unit (either ODFS III or Pace) to the dorsiflexors to treat foot drop for a period of 12 weeks.
  Interventions: Device: Functional Electrical Stimulation
- Ankle Foot Orthosis: The people in the Ankle Foot Orthosis group (AFO) will be asked to use their clinically prescribed AFO to treat drop foot for a period of 12 weeks.
  Interventions: Device: Ankle Foot Orthosis

INTERVENTIONS:
Device: Functional Electrical Stimulation
  Other Names: Odstock Dropped Foot Stimulator (ODFS) III; ODFS Pace
  Groups: Functional Electrical Stimulation
Device: Ankle Foot Orthosis
  Other Names: splint
  Groups: Ankle Foot Orthosis

SUMMARY:
This investigation consists of two parallel groups of participants who will follow the same protocol. The aim of the study is to investigate the effects of using Functional Electrical Stimulation/Ankle Foot Orthosis (AFO) or splint as an assistive mobility device over a 12 week period in people with MS who experience foot drop. Patients who are clinically prescribed FES will be invited to participate in the FES arm of the study. Patients who are clinically prescribed an AFO will be invited to participate in the AFO arm. Participants will be asked to make four visits to the gait laboratory at Queen Margaret University. Four weeks before the start of device use (Baseline - 4 weeks), start of device use (Baseline), after 6 weeks and 12 weeks of device use. Participants' walking will assessed using computerised three dimensional motion analysis, which will provide a detailed description of the movements (kinematics) of the lower limbs. Participants will also be asked to carry out a 10 metre walk and a two minute walk. Both gait analysis and the walking performance tests will be carried out with and without an assistive device; apart from their first session where participants will only be assessed without their assistive device.

Participants will be asked to wear an activity monitor for 7 days after each assessment. In addition participants will be asked to complete four short standardised questionnaires (MS walking scale, MS impact scale (MSIS-29), Fatigue severity score and the Leeds MS Quality of life score) at each assessment.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with Multiple Sclerosis
* Prescribed either AFO or FES to treat drop foot by their physiotherapist
* aged 18-75

Exclusion Criteria:

* Unable to walk 10 meters
* Bilateral device use
* Breastfeeding or pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Multiple Sclerosis who have been prescribed either FES or an AFO to treat foot drop by their physiotherapist.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in time taken for 10 meter walk test | change from baseline in 10m walk test at 12 weeks
  In the 10 meter walk test, the time taken by the participant to walk 10 meters is recorded. The test is repeated and the average is taken for analysis.

SECONDARY OUTCOMES:
Change in ankle dorsiflexion angle at initial contact | The change from baseline of the ankle dorsiflexion angle at initial contact from at 12 weeks
  The ankle dorsiflexion angle is derived from gait analysis. The angle of the ankle at the time the foot contacts the floor during a step is derived. This is repeated for at least 5 different walks, and the average of those 5 walks is calculated for further analysis.

OTHER OUTCOMES:
change in distance covered in two minutes | The change from baseline in the the 2 minute walk test at 12 weeks.
  During the 2 minute walk test the participant walks around an oval shaped track for 2 minutes. The distance covered in two minutes is taken for analysis.
The change in the MS walking scale (MSWS) | The change from baseline in the MSWS at 12 weeks
the change in the MS impact scale (MSIS29) | The change from basline in the MSIS29 at 12 weeks
The change in the Fatigue Severity Score (FSS) | The change from baseline in the FSS at 12 weeks
The change in the Leeds MS Quality of Life score (LMSQoL) | The change from baseline in the LMSQoL at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marietta L van der Linden, PhD, Principal Investigator — Queen Margaret University
Locations (1):
- Queen Margaret University, Musselburgh, East Lothian, United Kingdom

REFERENCES:
- [Derived] van der Linden ML, Hooper JE, Cowan P, Weller BB, Mercer TH. Habitual functional electrical stimulation therapy improves gait kinematics and walking performance, but not patient-reported functional outcomes, of people with multiple sclerosis who present with foot-drop. PLoS One. 2014 Aug 18;9(8):e103368. doi: 10.1371/journal.pone.0103368. eCollection 2014. PMID 25133535